CLINICAL TRIAL: NCT00545662
Title: Citicoline Brain Injury Treatment Trial
Brief Title: Study of Citicoline for the Treatment of Traumatic Brain Injury (COBRIT)
Acronym: COBRIT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Trial stopped due to futility.
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, William Friedewald, Professor, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BA-HD042; HD042687-04; HD042738-05; HD042678-03; HD042653-05; HD042689-05; HD042736-04; HD 042686-01A1; HD042652-04; HD042823-05
Record Dates: First submitted 2007-10-16; First posted 2007-10-17 (Estimated); Results first posted 2012-12-19 (Estimated); Last update posted 2012-12-19 (Estimated); Status verified 2012-11

CONDITIONS: Traumatic Brain Injury
Keywords: traumatic brain injury; cognition; behavioral outcome; functional outcome; treatment; early intervention; citicoline
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Cytidine Diphosphate Choline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Experimental): Placebo tablets formulated to resemble the citicoline treatment.
  Interventions: Drug: Placebo
- Citicoline (Experimental): Experimental treatment administered orally or enterally depending upon whether the participant can swallow at 1,000 mg twice a day for 90 days or until the 90-day outcome assessment.
  Interventions: Drug: citicoline

INTERVENTIONS:
Drug: Placebo — Drug Placebo Inactive twice a day given orally or enterally. The first dose is given within 24 hours of injury and treatment continues until 90 days or until the 90-day outcome assessment.
  Arms: Placebo
Drug: citicoline — 1000 mg twice a day orally or enterally. The first dose is within 24 hours of injury and treatment continues for 90-days or until the 90-day outcome assessment.
  Other Names: CDP-Choline, Cytidine 5-diphosphocholine, Somazina
  Arms: Citicoline

SUMMARY:
The Citicoline Brain Injury Treatment (COBRIT) is a randomized, double-blind, placebo controlled, multi-center trial of the effects of 90 days of citicoline on functional outcome in patients with complicated mild, moderate and severe traumatic brain injury.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) is a major cause of death and disability. In the United States alone approximately 1.4 million sustain a TBI each year, of which 50,000 people die, and over 200,000 are hospitalized. Despite numerous prior clinical trials no standard pharmacotherapy for the treatment of TBI has been established in either the acute or post acute setting. Citicoline is a naturally occurring endogenous compound. This compound offers the potential of employing neuroprotection, neuro-recovery and neurofacilitation to enhance recovery after TBI.

The primary goal of this study is to assess the efficacy of citicoline compared to placebo on functional and cognitive outcome in participants with traumatic brain injury.

ELIGIBILITY:
Inclusion Criteria:

1. Non-penetrating traumatic brain injury.
2. Age 18 (19 in Alabama) - 70 years.
3. GCS criteria on/off paralytics as specified in protocol
4. Reasonable expectation of completion of outcomes measures at a network center at six months post-injury.
5. Able to swallow oral medication or, if unable to swallow, a gastric tube or peg are placed by 23 hours after injury.
6. Reasonable expectation of enrollment within 24-hour time window.
7. English-speaking

Exclusion Criteria:

1. Intubated patients with GCS motor score = 6 and not meeting CT criteria.
2. Bilaterally fixed and dilated pupils
3. Positive pregnancy test, known pregnancy, or currently breast feeding
4. Evidence of diseases that interfere with outcome assessment
5. Current acetylcholinesterase inhibitor use (Appendix 1)
6. Imminent death or current life-threatening disease
7. Currently enrolled in another study
8. Prisoners

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1213 (Actual)
Dates: Start 2007-07; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherry Melton, MD, Principal Investigator — University of Alabama at Birmingham; Howard Eisenberg, MD, Principal Investigator — University of Maryland, Baltimore; Jack Jallo, MD, PhD, Principal Investigator — Temple University; Joseph Ricker, PhD, Principal Investigator — University of Pittsburgh; Shelly Timmons, MD, PhD, Principal Investigator — University of Tennessee Health Sciences Center; Ramon Diaz-Arrastia, MD, PhD, Principal Investigator — University of Texas Southwestern Medical Center; John Ward, MD, Principal Investigator — Virginia Commonwealth University; Nancy Temkin, PhD, Principal Investigator — University of Washington; Beth Ansel, PhD, Study Director — National Institute of Child Health and Human Development, National Center for Medical Rehabilitation Research; William Friedewald, MD, Principal Investigator — Columbia University Department of Biostatistics
Locations (8):
- United States (8):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Maryland, Baltimore, Baltimore, Maryland
  - Temple University, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Tennessee Health Sciences Center, Memphis, Tennessee
  - University of Texas, Southwestern Medical Center, Dallas, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Washington, Seattle, Washington

REFERENCES:
- [Derived] Zafonte RD, Bagiella E, Ansel BM, Novack TA, Friedewald WT, Hesdorffer DC, Timmons SD, Jallo J, Eisenberg H, Hart T, Ricker JH, Diaz-Arrastia R, Merchant RE, Temkin NR, Melton S, Dikmen SS. Effect of citicoline on functional and cognitive status among patients with traumatic brain injury: Citicoline Brain Injury Treatment Trial (COBRIT). JAMA. 2012 Nov 21;308(19):1993-2000. doi: 10.1001/jama.2012.13256. PMID 23168823

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant were recruited from eight level I trauma centers: Virginia Commonwealth University; University of Maryland; Temple University; University of Tennessee; University of Alabama (Birmingham); University of Texas Southwestern (Dallas); University of Pittsburgh; University of Washington. Recruitment began on 7/23/2007 and ended on 2/4/2011.
Groups:
- Control: The first dose of placebo was administered within 24 hours of traumatic brain injury. Placebo was administered orally or enterally depending upon whether the participant could swallow at 1,000 mg twice a day for 90 days or until the 90-day outcome assessment.
- Treatment: Treatment with citicoline begun within 24 hours of traumatic brain injury. Treatment was administered orally or enterally depending upon whether the participant could swallow at 1,000 mg twice a day for 90 days or until the 90-day outcome assessment.
Period: Overall Study
Arm/Group | Control | Treatment
Started | 606 | 607
Completed | 521 | 528
Not Completed | 85 | 79

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Treatment | Total
Number analyzed (Participants) | 606 | 607 | 1213
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 568 | 563 | 1131
  >=65 years | 38 | 43 | 81
Age Continuous [Mean (Standard Deviation); unit: years] | 41.1 (15.5) | 39.7 (16.2) | 40.4 (15.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 159 | 151 | 310
  Male | 447 | 456 | 903
Region of Enrollment [Number; unit: participants]
  United States | 606 | 607 | 1213

OUTCOME MEASURES:

1. Primary Outcome: Functional and Cognitive Outcome
Description: The primary outcome of this study was analyzed using a global statistic of the Network Core Battery. There were 9 scales: California Verbal Learning Test II (CVLT-II); Controlled Oral Word Association Test (COWAT); Digit Span (DS); Glasgow Outcome Scale Extended (GOSE); Processing Speed Index (PSI); Stroop Test 1 and 2 (ST1&2); and Trail Making Test part A and B (TMT parts A and B). Each scale was assigned cut-off for good outcome: GOSE>7, CVLT>36, PSI>85, TMT part A <42, TMT part B<138.1, DS>7.15, ST1<60.29, ST2<151.47, COWAT>32.5. Logistic regression was used to estimate the global OR.
Time Frame: 90 days
Population: The analysis included both the patients with complete outcome data and those with at least one measure. Patients who died were also included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Control | Treatment
Number analyzed (Participants) | 509 | 508
percentage of participants
  Glasgow Outcome Scale - Extended | 35.56 | 35.43
  California Verbal Learning Test | 60.48 | 57.71
  Processing Speed Index | 53.28 | 52.68
  Trail Making A | 61.96 | 64.96
  Trail Making B | 71.05 | 74.44
  Digit Span | 84.02 | 86.50
  Stroop Task 1 | 67.95 | 65.31
  Stroop Task 2 | 66.59 | 68.29
  Controlled Oral Word Association Test | 42.68 | 37.32
Statistical Analysis 1: Comparison: Control vs Treatment; Null hypothesis: The placebo and citicoline groups do not differ at 90-days on the Core Battery Power: 1. Two sided type I error of 0.05 2. 85% power 3. Expected OR=1.40 for the global statistic 4. Response rate in the control group 5. Correlations among the nine measures were accounted for. Response rates for the whole sample were a weighted average of the rates provided by TBI severity. 1240 participants were required to detect an OR >= 1.4 for the global statistic; Test type: Superiority or Other; p = 0.76, Regression, Logistic — a priori threshold for statistical significance is 0.05; Logistic regression estimated global OR. GEE accounted for correlations of the scales. Models adjusted for site & injury severity; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.83 to 1.14] — The odds in the citicoline group were compared to the odds in the placebo group

ADVERSE EVENTS:
Arm/Group | Control | Treatment
Serious Adverse Events (participants affected / at risk) | 117/606 | 117/607
Other Adverse Events (participants affected / at risk) | 452/606 | 449/607
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control (N=606) | Treatment (N=607)
CNS (Nervous system disorders) | 62 | 63
Cardiovascular (Vascular disorders) | 14 | 14
Respiratory (Respiratory, thoracic and mediastinal disorders) | 31 | 24
Dermatology/Skin (Skin and subcutaneous tissue disorders) | 3 | 1
Endocrine (Endocrine disorders) | 1 | 3
Digestive (Gastrointestinal disorders) | 7 | 13
Circulatory (Blood and lymphatic system disorders) | 6 | 11
Immune (Immune system disorders) | 5 | 4
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 5 | 5
Excretory/Urinary (Renal and urinary disorders) | 5 | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Control (N=606) | Treatment (N=607)
Gastrointestinal (Gastrointestinal disorders) | 184 | 193
Abnormal Lab (Investigations) | 143 | 175
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 157 | 132
Neurological (Nervous system disorders) | 319 | 308
Fever/Infection (Infections and infestations) | 118 | 127
Cardiovascular (Vascular disorders) | 88 | 86
Genitourinary (Renal and urinary disorders) | 73 | 75
Ophthalmologic (Eye disorders) | 51 | 48
Respiratory (Respiratory, thoracic and mediastinal disorders) | 132 | 143
Dermatologic/Skin (Skin and subcutaneous tissue disorders) | 69 | 59
Diaphoresis (General disorders) | 36 | 28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No